CLINICAL TRIAL: NCT05128045
Title: Weight Management & Wellness for People With Psychiatric Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Judith A. Cook, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-0118
Record Dates: First submitted 2021-10-20; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Obesity; Mental Illness
Keywords: Obesity, Weight Management, Serious Mental Illness
MeSH Terms: conditions — Obesity; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: NEW-R Intervention (Experimental): NEW-R Intervention plus services as usual
  Interventions: Behavioral: NEW-R
- Control (No Intervention): Services as usual

INTERVENTIONS:
Behavioral: NEW-R — Eight session class on nutrition, physical activity, diet, and weight management
  Arms: Experimental: NEW-R Intervention

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial to test the effectiveness of an intervention called Nutrition and Exercise for Wellness and Recovery (NEW-R) in promoting healthy eating and increased physical activity for better weight management among psychiatric outpatients.

DETAILED DESCRIPTION:
Weight management is a serious issue for individuals with mental health conditions, especially those who are taking psychiatric medications. The latest estimates are that over half of individuals receiving community mental health services are overweight or obese. This project's objective is to conduct a randomized controlled trial to test the effectiveness of an intervention called Nutrition and Exercise for Wellness and Recovery (NEW-R) in promoting healthy eating and increased physical activity for better weight management among psychiatric outpatients living and working in the community. It is an 8-week, recovery-oriented intervention that is co-led by a trained health educator and a certified mental health peer specialist. The study will take place at the UIC Department of Psychiatry in Chicago. Research participants will be recruited from the Department's outpatient clinics and other community programs, and randomly assigned to receive NEW-R along with services as usual or services as usual alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with a mental health disorder
* Patient of outpatient program
* Age 18 or older
* Being overweight or obese defined as BMI>=25
* Ability to understand spoken English

Exclusion Criteria:

* Residing in a nursing home
* Cardiac event in past 6 months
* Past episode of anorexia or bulimia
* Pregnancy
* Diagnosis with a terminal illness expected to result in death within 1 year
* Active alcohol or substance abuse or dependence
* Inability to provide informed consent due to diagnosis of dementia or cognitive impairment
* Inability to understand spoken English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Competence Scale from Baseline to 8-months | Study entry (Pre-intervention/T1), 2-months later (Post-Intervention 1/T2), & 6-months after T2 (Post-Intervention 2/T3
  Measures ability to stick with a weight management regimen and master new knowledge about diet and exercise. This 4-item scale using a 7-point Likert response format ranging from "not at all true" to "very true". The minimum value is 4 and the maximum is 28, with higher scores indicating a better outcome.
Change in Health Promoting Lifestyle Profile from Baseline to 8-months | Study entry (Pre-intervention/T1), 2-months later (Post-Intervention 1/T2), & 6-months after T2 (Post-Intervention 2/T3
  Measure of health promoting behavior. This is a 26-item scale with a 4-point Likert response format ranging from "never" to "routinely". Minimum value for this scale is 26 and the maximum is 104, with higher scores indicating a better outcome. The dimensions include nutrition, spirituality, and physical activity.

SECONDARY OUTCOMES:
Change in Self-Rated Abilities for Health Practices Scale from Baseline to 8-months | Study entry (Pre-intervention/T1), 2-months later (Post-Intervention 1/T2), & 6-months after T2 (Post-Intervention 2/T3
  Self perceived health management ability. This 7-item scale uses a 5-point Likert response format ranging from "not at all" to "completely". The minimum value is 7 and the maximum is 35, with higher scores indicating a better outcome.
Change in Weight from Baseline to 8-months | Study entry (Pre-intervention/T1), 2-months later (Post-Intervention 1/T2), & 6-months after T2 (Post-Intervention 2/T3
  Weight in pounds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brown C, Cook JA, Jonikas JA, Steigman PJ, Burke-Miller J, Hamilton MM, Rosen C, Tessman DC, Santos A. Nutrition and Exercise for Wellness and Recovery: A Randomized Controlled Trial of a Community-Based Health Intervention. Psychiatr Serv. 2023 May 1;74(5):463-471. doi: 10.1176/appi.ps.202200038. Epub 2022 Nov 15. PMID 36377367